CLINICAL TRIAL: NCT01716884
Title: China STEMI-PCI Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Abbott Medical Devices (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Yong Huo, Director of cardiovascular department, Peking University First Hospital
Other Study IDs: 2011[436]
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI; reperfution; primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. Registration
2. Performing in three stages
3. Major aim: Much more and standard reperfusion therapy in STEMI patients

ELIGIBILITY:
Inclusion Criteria:

* Onset of STEMI within 12h
* Onset of STEMI within 12-36h needing primary PCI

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI Patients enrolled and followed up 1 year
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The reperfusion ratio | up to 1 day

SECONDARY OUTCOMES:
Door to Balloon time | up to 1 day
BMS ratio | up to 1 day
health economic evaluation | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, China